CLINICAL TRIAL: NCT03980782
Title: The Effect of a Music Intervention on the Incidence, Severity and Duration of Delirium in Older Acute Care Patients
Brief Title: The Effect of Music Therapy on Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Mary Kovaleski, Principal Investigator, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-0319
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2019-12

CONDITIONS: Delirium
Keywords: Delirium elderly Music therapy; Elderly; Music Therapy
MeSH Terms: conditions — Delirium | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: A randomized control pilot study will be used to test the effect of a music therapist-developed, music listening intervention on delirium. Acutely ill patients will be randomized into a usual care control group or an experimental group receiving the music intervention twice daily for 30 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention (Experimental): Each participant will receive a 30 minute individual music intervention twice daily.
  Interventions: Other: Music Therapy
- Care as usual (No Intervention): Each participant will receive care as usual.

INTERVENTIONS:
Other: Music Therapy — Individualized music therapy developed playlist(s) that will be used based upon the latest Confusion Assessment Method result (hypoactive, hyperactive or no delirium) delivered twice daily.
  Arms: Music Intervention

SUMMARY:
The purpose of this study is to test the effect of a twice daily, 30-minute, interdisciplinary, music therapist developed, nurse initiated, music listening intervention on acutely ill older patients as compared to patients who receive care as usual. Half of the participants will receive music therapy and the other half will receive care as usual.

DETAILED DESCRIPTION:
Delirium is a complex, preventable, neuropsychiatric syndrome that is associated with higher mortality rates post discharge, increased hospital stays, increased mortality and an increased risk for developing dementia. Early, nonpharmacological treatment of delirium is preferable and supported by the literature to preserve patient safety. Music therapy is an evidence based, goal directed treatment process in which the music therapist and the patient maintain a state of well-being to achieve individualized patient goals. Music interventions are therapist developed and nurse initiated, in accordance to individual patient needs to maintain well-being, and show promise for improving attention and engagement. Understanding the effect of an individualized music intervention on the incidence, duration and severity of delirium has the potential to facilitate the use of cost-effective methods to modify individual environments to deliver appropriate care for acutely ill older adults. Purpose: The purpose of this study is to test the effect of an interdisciplinary music intervention on the incidence, severity and duration of delirium in older acutely ill adults. Methods: A randomized control pilot study will be used to test the effect of a music therapist-developed, music listening intervention on delirium. Acutely ill patients will be randomized into a usual care control group or an experimental group receiving the music intervention twice daily for 30 minutes. Data analysis: Descriptive statistics will be used to describe the sample. Independent t-tests will be used to examine group differences in delirium severity and duration. Chi-square analysis will be used to assess group differences in delirium incidence. Implications: For patients exposed to the stress of hospitalization, a music intervention may enhance delirium care and promote care that is safe and efficient.

ELIGIBILITY:
Inclusion Criteria:

Age 65 or older Admitted to the Progressive Care Unit (PCU), must be able to speak English Must be able to hear music through headphones. Must not have a documented history of dementia Must not have a documented history of permanent cognitive impairment, Must not be delirious at the beginning of the study (CAM negative) Must be able to sign a consent form.

Exclusion Criteria:

Age less than 65, Not admitted to the Progressive Care Unit, Positive for delirium (CAM positive) Does not speak English, Has a hearing impairment, Documented history of dementia Documented history of permanent cognitive decline Expected death within 24 hours of enrollment, Transferred off the floor Unable to sign consent.

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The effect of Music Therapy on the Incidence of Delirium in Older Acute Care Patients. | 2-3 months
  The incidence of delirium will be measured twice a day with the Confusion Assessment Method (CAM).

SECONDARY OUTCOMES:
The Effect of a Music Intervention on the Severity of Delirium in Older Acute Care Patients | 2-3 months
  The severity of Delirium will be determined using the Confusion Assessment Method- S (CAM-S assessment) twice a day once participants are CAM positive. The CAM-S, rate each symptom of delirium listed in the short CAM instrument as absent (0), mild (1), marked (2). Acute onset or fluctuation is rated as absent or present. Summarize these scores into a composite that ranges from 0-7 (higher scores indicate more severe delirium).

OTHER OUTCOMES:
The Effect of a Music Intervention on the Duration of Delirium in Older Acute Care Patients | 2-3 months
  Determine the duration of delirium will be determined by the number of days reporting a positive CAM...delirium resolution will be 48 hours without delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Spegman, PhD, Study Director — Geisinger Clinic
Locations (1):
- Geisinger CMC, Scranton, Pennsylvania, United States